CLINICAL TRIAL: NCT02434757
Title: Addition of H. P Acthar Gel to Treatment Regimen of Patients With Rheumatoid Arthritis Inadequately Controlled With Biologic Disease-Modifying Antirheumatic Drugs
Brief Title: Addition of H.P. Acthar Gel to Treatment Regimen of Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ronald J. Rapoport, MD (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Ronald J. Rapoport, MD, Ronald Jay Rapoport, MD, Phase III Clinical Research
Organization: Phase III Clinical Research (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT1
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acthar 40 U (Experimental): Acthar 40 U (0.5mL)
  Interventions: Drug: H.P. Acthar Gel

INTERVENTIONS:
Drug: H.P. Acthar Gel — Acthar 40 U given SC daily for 7 days. Depending on the response and the Investigator,Acthar 40 U will continue Acthar 40 U 2x per week or increase to Acthar 80 U daily for 7 days followed by 2x per week
  Other Names: Acthar; Repository Corticotropin Injection; ACTH Gel

SUMMARY:
This small study is to investigate the efficacy and safety of Acthar as an adjunct therapy in patients with active rheumatoid arthritis (RA) who have had an inadequate response to disease modifying antirheumatic drugs (DMARDs) and at least 3 biologic agents. An in adequate response is defined as having ≥ 6 tender joints, ≥ 6 swollen joints, plus C-Reactive Protein (CRP) levels and/or erythrocyte sedimentation rate (ESR) of ≥ 1.2 times the upper limit of normal in spite of aggressive treatment, including ≥ 7.5 mg/d prednisone. This will be a 20 week, prospective, multicenter, open-label study conducted at 3-4 university/medical centers and private practice settings in the US. A total of 20 eligible patients will be enrolled and other standard RA therapeutic agents, such as Methotrexate, DMARDs, non-steroidal anti-inflammatory drugs (NSAIDs), pain medications and others will not be discontinued. The primary endpoint will be the percentage of patients with reduction of ≥1.2 points of the Disease Activity Score in 28 joints (DAS-28) score.

DETAILED DESCRIPTION:
>

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of participation
* Have a confirmed diagnosis of RA based on the 2010 ACR/EULAR criteria
* Currently on aggressive treatment with an inadequate response or AE to stable dose of DMARDs and biologic agents for 3 months prior to screening, and stable doses of NSAIDs, prednisone or equivalent dose of corticosteroid (dose ≥7.5 mg/d), and analgesics for 28 days prior to screening. Have active RA, defined as ≥6 swollen joints, ≥6 tender joints, plus CRP levels an /or an ESR ≥1.2 the upper limit of normal
* RA for art least 24 months and receiving maximum tolerated doses of at lease 3 biologic agents (at least 1 of which is anti-TNF-a) for 3 months
* Tuberculosis has not occurred within the recent past, as proven by a conventional x-ray, negative tuberculosis shin test (PPD), or quantiferon gold

Exclusion Criteria:

* Presence of any condition which could confound interpretation of the data, such as inflammatory arthritis (eg. psoriatic arthritis, gout or pseudogout)
* Presence of systemic fungal infections, recent surgery (within prior 3 months), or active ulcer disease (within the past 5 years)
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic ,hematologic, gastrointestinal, pulmonary, cardiac, neurological or cerebral disease
* Have had in last three months or planning to receive live or live attenuated vaccines
* Concomitant medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in the study such as uncontrolled diabetes or hypertension
* History of or presence of active or latent tuberculosis (TB) based on QuantiFERON-TB gold test. Patients will be allowed in the study after receiving adequate treatment for TB
* Sensitivity to proteins of porcine origin
* History of cancer within the last 5 years, excluding basal cell carcinoma
* Glomerular filtration rate <30 mL/min -
* Uncontrolled diabetes mellitus
* Pregnant of lactating female patients. Each site to administer a pregnancy test to any female of childbearing potential before prescribing Acthar Gel. Only females with negative pregnancy test results are eligible. All sexually active males and females of childbearing potential must agree to use an adequate method of contraception throughout the period of the study.
* The following physical and laboratory test findings
* Patients with positive hepatitis B surface antigen
* Patients with positive hepatitis C antibody, who are also positive by recombinant immunoblot assay (RIBA) or by polymerase chain reaction (PCR)
* Hemoglobin level <8.5. g/dL
* White blood cell count <3000/mm (3 x 10/L)
* Serum Creatinine level >2 times upper limit of normal
* Serum alanine aminotransferase (ALT) or asparate amino- transferase (AST) >2 times upper limit of normal
* Any other laboratory test results that, in the opinion of the investigator might placed the patient at unacceptable risk for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with reduction of >1.2 points in DAS-28 score | After 12 weeks
20%, 50%, 70% Improvement based on American College of Rheumatology Criteria | After 12 weeks

SECONDARY OUTCOMES:
Improvement (decrease) in Vectra Disease Activity score | After 12 weeks
Improvement (decrease) in Health Assessment Questionnaire | After 12 weeks
Improvement in Functional Assessment of Chronic Illness Therapy Health Related Quality of Life Score | After 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Phase III Clinical Research, Fall River, Massachusetts, United States